CLINICAL TRIAL: NCT01832129
Title: Acceptance and Biomarker Response With Oral vs. Intramuscular Supplementation of Vitamin B12 in Primary Care
Brief Title: Vitamin B12 Acceptance and Biomarker Response Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other); Aarelab AG (Industry)
Responsible Party: Principal Investigator, Philipp Walter, PhD, MSc, University of Basel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PCRG_VB12_CM
Record Dates: First submitted 2013-04-05; First posted 2013-04-15 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Vitamin B 12 Deficiency
MeSH Terms: conditions — Vitamin B 12 Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- i.m. injection of Vitamin B12 (Active Comparator): Weekly i.m. injections of 1 mg Cyanocobolamin after 1, 2, and 3 weeks.
  Interventions: Drug: i.m. injection of vitamin B12
- Oral administration of vitamin B12 (Experimental): High dose (1 mg/day) oral Cyanocobolamin will be adminstrated with electronic adherence monitoring.
  Interventions: Drug: Oral administration of vitamin B12

INTERVENTIONS:
Drug: Oral administration of vitamin B12 — Daily high dose oral vitamin B12 (1mg) will be administered over 4 weeks. The patients adherence to this regimen will be monitored with an electronic punch card.
  Other Names: Cyanocobolamin; B12 "Ankermann" 1 mg
  Arms: Oral administration of vitamin B12
Drug: i.m. injection of vitamin B12 — Intramuscular injections of 1 mg vitamin B12 will be performed at days 7, 14, and 21.
  Other Names: Vitamin B12 intramuscular; Cyanocobolamin; Vitarubin Depot
  Arms: i.m. injection of Vitamin B12

SUMMARY:
In this study, biomarker response after supplementation with oral and intramuscular vitamin B12 will be compared in a randomized clinical trial. Electronic compliance monitoring will be used to control for non compliance as a possible confounder in oral treatment. Additionally subjective acceptance in terms of presumed preferences will be compared with oral vs. intramuscular supplementation of vitamin B12 in the view of the patient.

ELIGIBILITY:
Inclusion Criteria:

* General practitioner's prescription for Vitamin B12 deficiency testing
* Age> 18 years
* Ability to give written informed consent
* Vitamin B12 serum concentrations < 200pmol/l
* indication for vitamin B12 supplementation according to the General practitioners estimation

Exclusion Criteria:

* Patients with incorrect intake of vitamin preparations containing vitamin B12
* Patients with previously diagnosed dementia
* Patients with known hereditary transcobalamin transportation defects
* lack of written and/or oral understanding in German, French, Italian or English languages

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Biochemical response to vitamin B12 substitution | Day 28
  Vitamin B12 associated biomarkers (Vitamin B12, Holotranscobolamin, Homocystein, MCV, hypersegmentated neutrophils)

SECONDARY OUTCOMES:
taking and timing adherence with oral vitamin B12 | day 28
  Adherence to oral vitamin B12 supplementation will be measured with an electronic adherence monitoring device. The number of doses taken (taking adherence) and the number of doses taken within the defined time-frame (timing adherence) will be measured.
Comparison of patient acceptance of oral vs. i.m. vitamin B12 supplementation | day 0, day 28
  Acceptance of the two routes of administration of vitamin B12 substitution by the patients will be measured by specific questionnaires before and after exposure to the medication in both arms.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt E Hersberger, Professor, Study Chair — Pharmaceutical Care Research Group; Cyrill Jeger, MD, Principal Investigator; Philipp N Walter, MSc, Study Director — Pharmaceutical Care Research Group
Locations (1):
- Pharmaceutical Care Research Group, Basel, Basel, Switzerland

REFERENCES:
- [Derived] Metaxas C, Mathis D, Jeger C, Hersberger KE, Arnet I, Walter P. Early biomarker response and patient preferences to oral and intramuscular vitamin B12 substitution in primary care: a randomised parallel-group trial. Swiss Med Wkly. 2017 Apr 7;147:w14421. doi: 10.4414/smw.2017.14421. eCollection 2017. PMID 28421567